CLINICAL TRIAL: NCT06901648
Title: Efficacy and Safety of HS-20094, a Novel Dual GIP and GLP-1 Receptor Agonist, in Patients With Type 2 Diabetes: a Randomized, Placebo-controlled and Active Comparator-controlled Phase 2 Trial
Brief Title: A Study of HS-20094 in Patients With T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-20094-203
Record Dates: First submitted 2025-02-25; First posted 2025-03-30 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- HS-20094 5mg (Experimental)
  Interventions: Drug: HS-20094
- HS-20094 10mg (Experimental)
  Interventions: Drug: HS-20094
- HS-20094 15mg (Experimental)
  Interventions: Drug: HS-20094
- Dulaglutide 1.5mg (Active Comparator)
  Interventions: Drug: Dulaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Palcebo

INTERVENTIONS:
Drug: HS-20094 — Administrated by subcutaneous injection once a week
  Arms: HS-20094 10mg; HS-20094 15mg; HS-20094 5mg
Drug: Dulaglutide — Administrated by subcutaneous injection once a week
  Arms: Dulaglutide 1.5mg
Drug: Palcebo — Administrated by subcutaneous injection once a week
  Arms: Placebo

SUMMARY:
This is a 32-week, phase 2, randomized study, HS-20094 and placebo were double-blind, dulaglutide was open-label. Adults with T2D inadequately controlled with diet and exercise alone or with stable metformin, an HbA1c (glycated hemoglobin) ≥53 to ≤91 mmol/mol (≥7.0 % to≤10.5 %) were randomly assigned to receive 5 mg HS-20094, 10 mg HS-20094, 15 mg HS-20094, placebo, or 1.5 mg dulaglutide subcutaneously for 32 weeks. The primary endpoint was change in HbA1C from baseline to 32 weeks, and secondary endpoints included change in fasting glucose, body weight and several additional measures relevant for cardiovascular risks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 to 75 years of age, inclusive
2. Patients were diagnosed with T2DM for at least 3 months before screening.
3. Have an HbA1c value at screening of ≥7.0% and ≤10.5% and treated with diet and exercise alone or a stable dose of metformin (either immediate release or extended release, ≥1000mg/day and not more than the locally approved dose) for at least 2 months prior to screening
4. Body mass index (BMI）≥ 22 kg/m2.

Exclusion Criteria:

1. Type 1 diabetes, gestational diabetes, monogenic diabetes, secondary diabetes, or undetermined diabetes as assessed by the investigator
2. Acute or chronic pancreatitis at any time before screening, or serum lipase/amylase above the upper limit of normal at screening
3. A history of grade 3 hypoglycemia (hypoglycemia with a serious event of consciousness and/or physical alteration requiring assistance from another person for recovery) within 6 months before screening
4. Occurrence of diabetic ketoacidosis, hyperosmolar coma, or lactic acidosis two or more times within 6 months prior to screening
5. Occurrence of any of the following events within 6 months prior to screening: acute myocardial infarction, unstable angina, coronary artery bypass grafting, percutaneous coronary intervention (excluding diagnostic angiography), transient ischemic attack, cerebrovascular accident, decompensated congestive heart failure, or Class III or IV heart failure (NYHA classification)
6. Significant weight change (weight gain or loss ≥5%) within 3 months prior to screening (as reported by the participant)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
The change of HbA1c in the patients | From baseline to week 32

SECONDARY OUTCOMES:
The percentage of patients reaching the HbA1c target of ≤ 6.5% | From baseline to week 32
The percentage of patients reaching the HbA1c target of<7.0% | From baseline to week 32
The change in fasting blood glucose | From baseline to week 32
The change in C peptide | From baseline to week 32
The change of fasting insulin in the patients | From baseline to week 32
The change in body weight | From baseline to week 32
The percentage of patients with 5% or greater body weight loss | From baseline to week 32

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital (Zhu Xianyi Memorial Hospital), Tianjin, Tianjin Municipality, China